CLINICAL TRIAL: NCT00241397
Title: An Observational Study on the Presence of Depression and/or Anxiety Disorder in Patients Consulting the General Practitioner With Painful Physical Symptoms in Belgium and Luxemburg.
Brief Title: Study Evaluating Rhapsody Registry in Patients With Depression and Anxiety
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Other Study IDs: 0600B1-102003
Record Dates: First submitted 2005-10-17; First posted 2005-10-18 (Estimated); Last update posted 2007-03-15 (Estimated); Status verified 2007-03

CONDITIONS: Pain; Depression; Anxiety Disorder
Keywords: pain; depression; anxiety disorder
MeSH Terms: conditions — Pain; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of this study is to assess the prevalence of Major Depression and/or Anxiety Disorder in patients consulting the General Practitioner with acute or chronic painful physical symptoms and to identify risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient must be at least 18 years of age
* Consulting a General Practitioner for painful physical symptoms
* Written informed consent

Exclusion Criteria:

* Patient is unable to understand and comply with procedures of the study
* Patient is unable to complete the patient ratings
* Patient has an acute pain with an obvious cause

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2560
Dates: Start 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For Belgium, trials-BEL@wyeth.com
Locations (82):
- Belgium (82):
  - Aarschot
  - Aiseau-Presles
  - Anderlues
  - Andrimont
  - Angleur
  - Ans
  - Anthée
  - Auvelais
  - Avelgem
  - Beauraing
  - Beernem
  - Bekegem-Ichtegem
  - Belgrade
  - Bertogne
  - Betekom
  - Bierges
  - Binche
  - Bioul
  - Braine-l'Alleud
  - Bruges
  - Brussels
  - Charleroi
  - Ciney
  - Couillet
  - Deurne (Antwerpen)
  - Dworp
  - Eupen
  - Éghezée
  - Galmaarden
  - Goutroux
  - Grimminge
  - Hatrival
  - Hemiksem
  - Herenthout
  - Hoboken
  - Houdeng-Aimeries
  - Houdeng-Goegnies
  - Incourt
  - Itegem
  - Jabbeke
  - Jambes
  - Jodoigne
  - Kapellen
  - Kettenis
  - Klemskerke
  - Kuurne
  - Laarne
  - Lasne
  - Leuven
  - Lobbes
  - Luttre
  - Merksem
  - Mélin
  - Monceau-sur-Sambre
  - Morlanwelz-Mariemont
  - Moustier S/S
  - Noorderwijk
  - Oudenaarde
  - Ranst
  - Rèves
  - Rixensart
  - Romsée
  - Rotselaar
  - Ruddervoorde
  - Sainte-Marie-sur-Semois
  - Schildewindeke
  - Schoten
  - St-Joris Winge
  - Steenokkerzeel
  - Waarschoot
  - Waha
  - Walem
  - Wavre
  - Wetteren
  - Wevelgem
  - Wilrijk
  - Wommelgem
  - Wondelgem
  - Wuustwezel-Gooreind
  - Zelzate
  - Zemst
  - Zétrud-Lumay